CLINICAL TRIAL: NCT04739397
Title: Evaluation of the EpiGlare Tester for the Measurement of Glare-Induced Changes in BSCVA in Subjects With and Without Cataracts
Status: Completed | Type: Observational
Sponsor: Epico, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: EG-001
Record Dates: First submitted 2016-01-25; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2016-01

CONDITIONS: Cataract
Keywords: Disability glare; contrast sensitivity; cataract; method evaluation; glare test
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cataract: Patients with bilateral cataracts with Lens grade 2+ or greater, cataract classification nuclear, cortical or posterior subcapsular
  Interventions: Device: Glare Testing
- Non-Cataract: patients with bilateral clear lenses (no cataracts)
  Interventions: Device: Glare Testing

INTERVENTIONS:
Device: Glare Testing — Vision in Cataract patients were tested with and without the EpiGlare Tester
  Other Names: EpiGlare Tester

SUMMARY:
The EpiGlare Tester will identify visual disability resulting from the glare experienced by subjects with cataracts in the glare-induced change in best spectacle corrected visual acuity (BSCVA).

DETAILED DESCRIPTION:
Inclusion Criteria:

1. Are 18 years of age or older.
2. Have been evaluated by an opthalmologist and have a lens determination of either Normal or Cataract in each eye based on slit lamp examination.

   1. Normal = lens opacity of clear or trace
   2. Cataract = lens opacity of 2+ or greater
3. Have written informed consent as required by the site's IRB and received a copy.
4. Are willing and able to comply with testing according to the Investigator.

Exclusion Criteria:

1. Best corrected visual acuity is worse than 20/60 in either eye
2. Have occular pathology including corneal or macular disease or advanced glaucoma
3. Have cognitive dysfunction which limits the ability to cooperate with testing.
4. Have presence or history of any other condition or finding or concomitant medication that, in the investigator's opinion, makes the subject unsuitable as a candidate for EpiGlare or study participation or may confound the outcome of the study.

ELIGIBILITY:
Inclusion Criteria:

clear lenses OU cataracts OU willing to comply with testing

Exclusion Criteria:

BCVA < 20/63 either eye ocular pathology (ie corneal, macular disease, advanced glaucoma) cognitive dysfunction other conditions that in the investigators opinion made the subject unsuitable candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Candidates were identified from the investigator's usual clinic population. Subjects presenting to the investigators clinic were examined according to the usual procedures. Subjects were classified as having either bilateral cataracts or clear lenses in both eyes
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change in best spectacle corrected visual acuity (BSCVA) measurements before and after glare testing using the EpiGlare Tester as the glare source. | up to 16 months
  Change in best spectacle corrected visual acuity (BSCVA) measurements before and after glare testing using the EpiGlare Tester as the glare source in patients with and without cataracts.

SECONDARY OUTCOMES:
Evaluation of functional visual ability using driving and glare subscales from the Refractive Status Vision Profile (RSVP) questionnaire | up to 16 months
  Correlation of the EpiGlare Tester's glare-induced changes in BSCVA with functional glare disability, as measured by the glare subcategory from the RSVP questionnaire

OTHER OUTCOMES:
User's assessment using a subjective questionnaire. | up to 16 months
  Users evaluated the device using a subjective questionnair

CONTACTS AND LOCATIONS:
Overall Officials: Nicole R Fram, MD, Principal Investigator — Advanced Vision Care; Samuel Masket, MD, Principal Investigator — Advanced Vision Care; Fancis W Price, MD, Principal Investigator — Price Vision Group; R. Doyle Stulting, MD, PhD, Principal Investigator — Woolfson Eye Institute
Locations (1):
- The Eye Center of Columbus, Columbus, Ohio, United States

REFERENCES:
- [Background] Epitropoulos AT, Fram NR, Masket S, Price FW Jr, Snyder ME, Stulting RD. Evaluation of a New Controlled Point Source LED Glare Tester for Disability Glare Detection in Participants With and Without Cataracts. J Refract Surg. 2015 Mar;31(3):196-201. doi: 10.3928/1081597X-20150225-03. PMID 25751837